CLINICAL TRIAL: NCT04715035
Title: Efficacy of Eccentric Exercises in Individuals With Frozen Shoulder: A Randomized Controlled Clinical Trial
Brief Title: Efficacy of Eccentric Exercises in Individuals With Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Durand, Argentina (Other)
Responsible Party: Principal Investigator, Pablo Policastro, Physical Therapy, Hospital Durand, Argentina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Policastro.ECA.HombroCongelado
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Frozen Shoulder; Capsulitis, Adhesive; Capsulitis of Shoulder
Keywords: frozen shoulder; eccentric exercise; rehabilitation; physical therapy
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (Active Comparator): Physical therapy: education, mobilizations, stretch, active exercises, home excercises.
  Interventions: Other: Physical therapy interventions
- Conventional treatment + eccentric exercises (Experimental): Physical therapy: education, mobilizations, stretch, active exercises, home exercises, eccentric exercises.
  Interventions: Other: Physical therapy interventions

INTERVENTIONS:
Other: Physical therapy interventions — mobilization, stretch, education, eccentric exercises

SUMMARY:
Frozen shoulder is a musculoskeletal condition with a strong negative impact on activities of daily living, producing pain, disability, anxiety, and sleep disorders. It has a worldwide prevalence of 5.3%, increasing from 10 to 38% in patients with diabetes and thyroid conditions. This clinical entity manifests itself mainly in women between 40 and 65 years of age. Its resolution time is long and can reach 42 months with symptoms that persist throughout life.

In the clinical evaluation, patients with Frozen Shoulder are manifested mainly by presenting mobility deficits. Previous studies described different structural alterations that may justify this clinical condition and its consequences, such as, for example, fibrosis of the coracohumeral ligament, alterations of the rotator interval, and of the axillary recess.

Although passive structures are believed to be primarily involved in this condition, A series of five cases in which patients with frozen shoulder presented a significant increase in mobility after a general anesthetic block. The data obtained from this study and the different complications presented by patients with CH suggest that it is necessary to further understand the role of the rotator cuff in this clinical condition.

Eccentric exercises consist of contracting the muscle to control or decelerate a load while the muscle or tendon is lengthening or remaining stretched. This intervention has been proposed for the treatment of tendinopathies in different body regions.

DETAILED DESCRIPTION:
A randomized controlled clinical trial with two parallel groups will be carried out. Evaluators will be blinded to the treatment group and therapists will be unique to each group. This study will follow the CONSORT guidelines.

Randomization by blocks between groups will be carried out through the website www.randomization.com and the sequence will be stored in sealed and opaque envelopes to maintain allocation confidentiality. This process will be carried out by an independent researcher, who will not be involved in the assessment and treatment. The allocation of subjects will be revealed to the researcher responsible for the treatment by opening the envelope before the start of the intervention. The researcher responsible for the evaluation will be blinded to the treatment group. The individuals will be blinded in relation to the study hypothesis and will not have contact with the participants of the same or the other group.

Initially, all participants will undergo screening to assess the inclusion and non-inclusion criteria of the study. All individuals who meet the eligibility criteria will undergo an anamnesis to collect personal, sociodemographic, pain history, and primary and secondary outcomes measurements.

ELIGIBILITY:
Inclusion Criteria:

* History of diffuse-onset shoulder pain of at least one month
* Gradual loss of passive external rotation of at least 50% compared to the contralateral side

Exclusion Criteria:

- History of shoulder fracture/ surgery

* Shoulder pain reproduced by passive movement of the cervical spine
* History of rheumatoid arthritis
* Shoulder immobilization for more than 5 days
* Bilateral frozen shoulder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Shoulder Function | From enrollment to the end of treatment at 12 weeks. In the follow-up at 3 months and 9 months from the end of treatment.
  American Shoulder and Elbow Surgeons scale (ASES). This scale has a score between 0 to 100. When the score is more close to 0 Worst is the function of the shoulder and when is approximate 100, it is better.

SECONDARY OUTCOMES:
Range of Movement | From enrollment to the end of treatment at 12 weeks. In the follow-up at 3 months and 9 months from the end of treatment.
  An inclinometer will assess flexion, external rotation, and internal rotation range of movement. The higher the value, the better.
Perceived Pain | From enrollment to the end of treatment at 12 weeks. In the follow-up at 3 months and 9 months from the end of treatment.
  The perceived pain is going to be assessed by a Visual Analogue Scale from 0 to 10, where the score close to 0 is worst, and approximate to 10 is better.
Pennation Angle | From enrollment to the end of treatment at 12 weeks. In the follow-up at 3 months and 9 months from the end of treatment.
  It is going to be assessed by an ultrasound device
Fear avoidance | From enrollment to the end of treatment at 12 weeks. In the follow-up at 3 months and 9 months from the end of treatment.
  Fear Avoidance Beliefs Questionnaire This scale has a score between 0 to 96. When the score is more close to 96 worst is the fear avoidance and when is approximate to 0, it is better.
Perceived Quality of life | From enrollment to the end of treatment at 12 weeks. In the follow-up at 3 months and 9 months from the end of treatment.
  European Quality of Life Scale of five domains (EQ5D-3L). This scale has five items with a score between 1 to 3. When the score is more close to 3 worst is the quality of life and when is approximate to 1, it is better in each item. Also has a visual analogue scale of 100 points to assess the health condition, when the score is more close to 0 worst is the quality of life and when is approximate to 100 it is better.
Muscle Thickness | From enrollment to the end of treatment at 12 weeks. In the follow-up at 3 months and 9 months from the end of treatment.
  It is going to be assessed by an ultrasound device
Pain Catastrophizing | From enrollment to the end of treatment at 12 weeks. In the follow-up at 3 months and 9 months from the end of treatment.
  Pain Catastrophizing Scale (PCS)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Camargo, PhD, Study Director — University of São Carlos
Locations (1):
- Durand Hospital, Buenos Aires, Buenos Aires City, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Ryan V, Brown H, Minns Lowe CJ, Lewis JS. The pathophysiology associated with primary (idiopathic) frozen shoulder: A systematic review. BMC Musculoskelet Disord. 2016 Aug 15;17(1):340. 2. Kelley MJ, McClure PW, Leggin BG. Frozen shoulder: evidence and a proposed model guiding rehabilitation. J Orthop Sports Phys Ther. 2009 Feb;39(2):135-48. 3. Lewis J. Frozen shoulder contracture syndrome - Aetiology, diagnosis and management. Man Ther. 2015 Feb;20(1):2-9. 4. Chan HBY, Pua PY, How CH. Physical therapy in the management of frozen shoulder. Singapore Med J. 2017 Dec;58(12):685-689. 5. Kelley MJ, Shaffer MA, Kuhn JE, Michener LA, Seitz AL, Uhl TL, Godges JJ, McClure PW. Shoulder pain and mobility deficits: adhesive capsulitis. J Orthop Sports Phys Ther. 2013 May;43(5):A1-31. 6. Hollmann L, Halaki M, Kamper SJ, Haber M, Ginn KA. Does muscle guarding play a role in range of motion loss in patients with frozen shoulder? Musculoskelet Sci Pract. 2018 Oct;37:64-68.